CLINICAL TRIAL: NCT04970381
Title: An Exploratory Study of Effectiveness and Safety of Rivaroxaban in Patients With Left Ventricular Thrombus
Brief Title: An Exploratory stuDy of effectIveneSs and Safety of rivarOxaban in Patients With Left VEntricular Thrombus (R-DISSOLVE)
Acronym: R-DISSOLVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FW-2020-1380
Record Dates: First submitted 2021-07-11; First posted 2021-07-21 (Actual); Results first posted 2024-08-02 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-02

CONDITIONS: Ventricular Mural Thrombosis
MeSH Terms: interventions — Rivaroxaban

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rivaroxaban (Experimental): Rivaroxaban: Patients with ventricular mural thrombus in the study receive rivaroxaban anticoagulant therapy for 12 weeks. The dosage of rivaroxaban was typically 20mg once daily, or 15mg once daily if patients were on dual antiplateletagents, or with creatinine clearance of 30-50mL/min.
  Interventions: Drug: Rivaroxaban

INTERVENTIONS:
Drug: Rivaroxaban — Rivaroxaban: Patients with ventricular mural thrombus in the study receive rivaroxaban anticoagulant therapy for 12 weeks. The dosage of rivaroxaban was typically 20mg once daily, or 15mg once daily if patients were on dual antiplateletagents, or with creatinine clearance of 30-50mL/min.

SUMMARY:
To study the effect of rivaroxaban anticoagulant therapy for 12 weeks in patients with left ventricular mural thrombus by contrast echocardiography before and after treatment, so as to provide basis and foundation for further study and treatment selection in the future; To provide further relevant data for the treatment outcome, treatment duration and influencing factors of left ventricular mural thrombosis; It is of great sociological and health economic significance to find more effective and safe anticoagulant treatment strategies for patients with left ventricular mural thrombosis, which will reduce the incidence of embolism and bleeding.

ELIGIBILITY:
Inclusion Criteria:

1. Patients over 18 years old;
2. Patients with left ventricular thrombus newly found by body surface ultrasound less than or equal to 3 months before selection, with no limitation on basic diseases;
3. Patients who received standard anticoagulant therapy for less than 4 weeks before enrollment did not use antiplatelet drugs or only used single antiplatelet drugs;
4. The patients voluntarily joined the study and signed the informed consent.

Exclusion Criteria:

1. Patients with contraindications to rivaroxaban anticoagulation therapy;
2. Patients with a history of acute pulmonary embolism or deep venous thrombosis within a week need intensive anticoagulant therapy;
3. Patients with history of hemorrhagic stroke within one week;
4. Patients with cardiac benign and malignant tumors;
5. Aspirin and P2Y12 receptor antagonists should be kept;
6. In patients with severe hepatic and renal insufficiency, alanine aminotransferase > 3 times the upper limit and total bilirubin > 2 times the upper limit, creatinine clearance rate < 15ml / min / 1.73m2;
7. The patient's history of intracerebral hemorrhage and active hemorrhage was 8 months;
8. Patients with hematological diseases, hemoglobin < 100g / L, platelet < 80 x 10^9 / L;
9. Women with pregnancy status, planned pregnancy and lactation period;
10. Patients with life expectancy less than 1 year;
11. Patients enrolled in other clinical studies;
12. Other situations considered unsuitable by the researcher. Note: anticoagulant therapy can be given to patients with left ventricular thrombosis combined with hemorrhagic stroke ≥ 4 weeks or recent ischemic stroke / transient ischemic attack according to the specific situation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2020-09-27 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-10-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai Hospital, Chinese Academy of Medical Sciences & Pecking Union Medical College, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lee JM, Park JJ, Jung HW, Cho YS, Oh IY, Yoon CH, Suh JW, Chun EJ, Choi SI, Youn TJ, Lim C, Cho GY, Chae IH, Park KH, Choi DJ. Left ventricular thrombus and subsequent thromboembolism, comparison of anticoagulation, surgical removal, and antiplatelet agents. J Atheroscler Thromb. 2013;20(1):73-93. doi: 10.5551/jat.13540. Epub 2012 Sep 18. PMID 22986555
- [Background] O'Gara PT, Kushner FG, Ascheim DD, Casey DE Jr, Chung MK, de Lemos JA, Ettinger SM, Fang JC, Fesmire FM, Franklin BA, Granger CB, Krumholz HM, Linderbaum JA, Morrow DA, Newby LK, Ornato JP, Ou N, Radford MJ, Tamis-Holland JE, Tommaso CL, Tracy CM, Woo YJ, Zhao DX, Anderson JL, Jacobs AK, Halperin JL, Albert NM, Brindis RG, Creager MA, DeMets D, Guyton RA, Hochman JS, Kovacs RJ, Kushner FG, Ohman EM, Stevenson WG, Yancy CW; American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines. 2013 ACCF/AHA guideline for the management of ST-elevation myocardial infarction: a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines. Circulation. 2013 Jan 29;127(4):e362-425. doi: 10.1161/CIR.0b013e3182742cf6. Epub 2012 Dec 17. No abstract available. PMID 23247304
- [Background] Ibanez B, James S, Agewall S, Antunes MJ, Bucciarelli-Ducci C, Bueno H, Caforio ALP, Crea F, Goudevenos JA, Halvorsen S, Hindricks G, Kastrati A, Lenzen MJ, Prescott E, Roffi M, Valgimigli M, Varenhorst C, Vranckx P, Widimsky P; ESC Scientific Document Group. 2017 ESC Guidelines for the management of acute myocardial infarction in patients presenting with ST-segment elevation: The Task Force for the management of acute myocardial infarction in patients presenting with ST-segment elevation of the European Society of Cardiology (ESC). Eur Heart J. 2018 Jan 7;39(2):119-177. doi: 10.1093/eurheartj/ehx393. No abstract available. PMID 28886621
- [Background] Schulman S, Kearon C; Subcommittee on Control of Anticoagulation of the Scientific and Standardization Committee of the International Society on Thrombosis and Haemostasis. Definition of major bleeding in clinical investigations of antihemostatic medicinal products in non-surgical patients. J Thromb Haemost. 2005 Apr;3(4):692-4. doi: 10.1111/j.1538-7836.2005.01204.x. PMID 15842354
- [Background] Eikelboom JW, Connolly SJ, Bosch J, Dagenais GR, Hart RG, Shestakovska O, Diaz R, Alings M, Lonn EM, Anand SS, Widimsky P, Hori M, Avezum A, Piegas LS, Branch KRH, Probstfield J, Bhatt DL, Zhu J, Liang Y, Maggioni AP, Lopez-Jaramillo P, O'Donnell M, Kakkar AK, Fox KAA, Parkhomenko AN, Ertl G, Stork S, Keltai M, Ryden L, Pogosova N, Dans AL, Lanas F, Commerford PJ, Torp-Pedersen C, Guzik TJ, Verhamme PB, Vinereanu D, Kim JH, Tonkin AM, Lewis BS, Felix C, Yusoff K, Steg PG, Metsarinne KP, Cook Bruns N, Misselwitz F, Chen E, Leong D, Yusuf S; COMPASS Investigators. Rivaroxaban with or without Aspirin in Stable Cardiovascular Disease. N Engl J Med. 2017 Oct 5;377(14):1319-1330. doi: 10.1056/NEJMoa1709118. Epub 2017 Aug 27. PMID 28844192
- [Background] Lip GY, Hammerstingl C, Marin F, Cappato R, Meng IL, Kirsch B, van Eickels M, Cohen A; X-TRA study and CLOT-AF registry investigators. Left atrial thrombus resolution in atrial fibrillation or flutter: Results of a prospective study with rivaroxaban (X-TRA) and a retrospective observational registry providing baseline data (CLOT-AF). Am Heart J. 2016 Aug;178:126-34. doi: 10.1016/j.ahj.2016.05.007. Epub 2016 May 17. PMID 27502860
- [Derived] Yang Q, Quan X, Zhang Y, Feng G, Zhang T, Wang C, Yu D, Yu L, Yang Y, Zhu J, Liang Y. An exploratory study of effectiveness and safety of rivaroxaban in patients with left ventricular thrombus (R-DISSOLVE). J Thromb Thrombolysis. 2023 May;55(4):649-659. doi: 10.1007/s11239-023-02790-1. Epub 2023 Mar 20. PMID 36940069

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rivaroxaban
Started | 75
Completed | 66
Not Completed | 9

BASELINE CHARACTERISTICS:
Groups:
- Rivaroxaban: Rivaroxaban: Patients with ventricular mural thrombus in the study receive rivaroxaban anticoagulant therapy for 12 weeks
Arm/Group | Rivaroxaban
Number analyzed (Participants) | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.3 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 64
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 75
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  China | 75
BMI, kg/m2 [Mean (Standard Deviation); unit: kg/m2] | 24.5 (3.1)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Left Ventricular Thrombus Resolution at 12 Weeks/Number of Participants at 12 Weeks
Description: the rate of left ventricular thrombus resolution at 12 weeks=Number of Participants with left ventricular thrombus resolution at 12 weeks/Number of Participants at 12 weeks
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Rivaroxaban
Number analyzed (Participants) | 64
Participants | 50

2. Secondary Outcome: Number of Participants With Left Ventricular Thrombus Resolution at 6 Weeks/Number of Participants at 6 Weeks
Description: The left ventricular thrombus resolution rate at 6 weeks=Number of Participants With Left Ventricular Thrombus Resolution at 6 Weeks/Number of Participants at 6 Weeks
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Rivaroxaban
Number analyzed (Participants) | 62
Participants | 41

3. Secondary Outcome: Number of Participants With Left Ventricular Thrombus Resolution or Reduction at 6 Weeks/Number of Participants at 6 Weeks
Description: The left ventricular thrombus resolution or reduction rate at 6 weeks=Number of Participants With Left Ventricular Thrombus Resolution or reduction at 6 Weeks/Number of Participants at 6 Weeks
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Rivaroxaban
Number analyzed (Participants) | 62
Participants | 59

4. Secondary Outcome: Number of Participants With Left Ventricular Thrombus Resolution or Reduction at 12 Weeks/Number of Participants at 12 Weeks
Description: The left ventricular thrombus resolution or reduction rate at 12 weeks=Number of Participants With Left Ventricular Thrombus Resolution or reduction at 12 Weeks/Number of Participants at 12 Weeks
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Rivaroxaban
Number analyzed (Participants) | 64
Participants | 61

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Rivaroxaban
All-Cause Mortality (participants affected / at risk) | 2/75
Serious Adverse Events (participants affected / at risk) | 7/75
Other Adverse Events (participants affected / at risk) | 1/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rivaroxaban (N=75)
Rehospitalization (Cardiac disorders) | 7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rivaroxaban (N=75)
Allergy causing rivaroxaban discontinuation (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-09-10): https://cdn.clinicaltrials.gov/large-docs/81/NCT04970381/Prot_SAP_000.pdf
  • Informed Consent Form (2020-09-10): https://cdn.clinicaltrials.gov/large-docs/81/NCT04970381/ICF_001.pdf